CLINICAL TRIAL: NCT00079495
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability and Efficacy of NBI-5788 in Patients With Relapsing Multiple Sclerosis
Brief Title: Evaluation of an Altered Peptide Ligand (NBI-5788) in Patients With Relapsing Multiple Sclerosis (MS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Collaborators: Immune Tolerance Network (ITN) (Network)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NBI-5788-0201; MS APL; Neurocrine
Record Dates: First submitted 2004-03-08; First posted 2004-03-10 (Estimated); Last update posted 2008-03-21 (Estimated); Status verified 2007-09

CONDITIONS: Multiple Sclerosis
Keywords: MS; Autoimmune disease; relapsing; progressive; Myelin; Myelin Basic Protein; MBP; acute fulminating; chronic progressive; Altered Peptide Ligand; APL; Neurocrine; NBI-5788; Relapse
MeSH Terms: conditions — Multiple Sclerosis; Autoimmune Diseases; Recurrence | interventions — NBI 5788

INTERVENTIONS:
Drug: NBI-5788

SUMMARY:
We are studying this investigational drug treatment, comparing it with placebo, to evaluate whether it is effective in reducing the number of MRI lesions with a minimum number of side effects. The investigational drug will be administered in the clinic weekly for 5 injections (induction phase) then monthly for 8 additional injections (maintenance phase).

Approximately 150 male and female patients (100 active and 50 placebo), aged 18 to 55 years, with relapsing MS and at least one but no more than 10 total Gd-enhancing lesions on cranial MRI scans during the run-in phase will be randomized into this study.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled trial in which qualifying patients will be randomized 2:1 to receive active drug or placebo. Eligible patients must have MS with relapse, have had one or more relapses during the prior 2 years, 1-10 gadolinium (Gd)-enhancing lesions on the Run-in MRI, and an EDSS of 6.5 or less. There are exclusions for certain prior MS treatments and medical / psychiatric conditions. Following a 4-week run-in phase in which patients will have a baseline MRI, patients will enter a 4 week induction phase, during which they will be receive injections weekly (5 doses), then a 32-week maintenance phase during which injections are monthly (8 doses). A final follow-up visit will be conducted 4 weeks after the last injection. The primary efficacy parameter is a summary change score of the mean number of total Gd-enhancing lesions at weeks 36 and 40 minus the mean number for the two baseline scans. Safety monitoring will include AE/SAE reporting, physical exams, vital signs, ECG. CXR, laboratory tests, neurologic evaluations, and systemic hypersensitivity and injection site assessments. All study medications will be administered by study personnel and patients will remain under observation for a minimum of 2 hours post-injection. An independent Data Safety and Monitoring Board will oversee the safety of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 55 years of age
* Diagnosed with relapsing multiple sclerosis, with at least one relapse in the last two years
* Females must not plan on becoming pregnant
* Females must either be post-menopausal, surgically incapable of bearing children, or practicing an acceptable method of birth control and willing to continue birth control until 30 days after the last dose of study drug
* Males must not intend to impregnate a partner during the study or for 30 days after the study and must also practice acceptable birth control with their partners

Exclusion Criteria:

* Significant long-lasting disease of the immune system other than multiple sclerosis
* Past or current medical disease (heart, liver, kidney, etc.) including severe asthma, cancer or advancing brain or spinal cord disorder
* Known or suspected long-lasting infectious disease including HIV, hepatitis B, or hepatitis C
* Treatment with certain steroid or hormone medications within 30 days before the pre-study MRI scan
* Treatment with other medications that suppress the immune system within 6 months before the pre-study MRI scan
* Certain treatments and medications are not allowed
* Laboratory and other tests will be performed to determine further eligibility
* History of drug or alcohol abuse in the last year
* History of medical or psychiatric condition that could pose a risk for participation in the study
* Females who are pregnant or breast feeding
* Participation in any other trial of an investigational agent within 90 days before the start of the study
* History of not following instructions with past therapy.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150
Dates: Start 2003-07; Study Completion 2005-04

CONTACTS AND LOCATIONS:
Overall Officials: Chris O'Brien, MD, Study Director — Neurocrine Biosciences